CLINICAL TRIAL: NCT02679092
Title: Mifepristone Versus Osmotic Dilators in Conjunction With Misoprostol for Cervical Preparation Prior to D&E at 14-19 Weeks
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding changes.
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-36302
Record Dates: First submitted 2016-02-03; First posted 2016-02-10 (Estimated); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Legally Induced Abortion Without Mention of Complication
Keywords: Induced Abortion; Mifepristone; Dilation and Evacuation; Cervical Preparation; Osmotic Dilators; Misoprostol
MeSH Terms: conditions — Dilatation, Pathologic | interventions — Misoprostol; Mifepristone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Dilapan (14wks 0days-15wks, 6days) (Active Comparator): The clinician will place 1 to 2 osmotic cervical dilators (Dilapan-S) (4mm x 65mm) the day before the participant's procedure.
  Interventions: Device: Hygroscopic cervical dilators
- Dilapan (16wks 0days-18wks, 6days) (Active Comparator): The clinician will place 3 to 5 osmotic cervical dilators (Dilapan-S) (4mm x 65mm). Patients in this arm will also receive 200 mg misoprostol PO 30-90 minutes prior to their procedure.
  Interventions: Drug: Misoprostol; Device: Hygroscopic cervical dilators
- Mifepristone (14wks 0days-15wks, 6days) (Experimental): The patient will be administered mifepristone (200mg) orally with juice or water by the clinician or study investigator. Patients in this arm will also receive 200 mg misoprostol PO 30-90 minutes prior to their procedure.
  Interventions: Drug: Misoprostol; Drug: Mifepristone
- Mifepristone (16wks 0days-18wks, 6days) (Experimental): The patient will be administered mifepristone (200mg) orally with juice or water by the clinician or study investigator. Patients in this arm will also receive 200 mg misoprostol PO 30-90 minutes prior to their procedure.
  Interventions: Drug: Misoprostol; Drug: Mifepristone

INTERVENTIONS:
Drug: Misoprostol — 400 mcg buccal 60-90 minutes prior to procedure
  Other Names: Cytotec
  Arms: Dilapan (16wks 0days-18wks, 6days); Mifepristone (14wks 0days-15wks, 6days); Mifepristone (16wks 0days-18wks, 6days)
Drug: Mifepristone — 200 mg PO on the day prior to D&E
  Other Names: Danco; Mifeprex
  Arms: Mifepristone (14wks 0days-15wks, 6days); Mifepristone (16wks 0days-18wks, 6days)
Device: Hygroscopic cervical dilators — osmotic cervical dilators inserted through the internal os
  Other Names: Dilapan-S
  Arms: Dilapan (14wks 0days-15wks, 6days); Dilapan (16wks 0days-18wks, 6days)

SUMMARY:
Dilation and evacuation (D&E) is a common surgical procedure in the U.S. Adequate pre-operative preparation of the uterine cervix is an important part of preventing complications of the procedure. Traditionally, the uterine cervix is prepared for the procedure using water-attracting dilators, which are placed via a speculum exam and cause discomfort for many women. The objective of this study is to investigate the comparative effectiveness of mifepristone (an oral tablet) versus dilators for cervical preparation for D&E.

ELIGIBILITY:
Inclusion Criteria:

* >18 Years Old
* Viable, Singleton pregnancy
* Voluntarily seeking abortion between 14-19 weeks gestation
* Able to give informed consent and comply with study protocol
* Fluent in English or Spanish

Exclusion Criteria:

* Allergy to study drugs

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-04 (Estimated); Primary Completion 2020-02 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Procedure Time | Intraoperative
  Measured as time from speculum insertion to removal.

SECONDARY OUTCOMES:
Cervical Dilation | Baseline
  Measured by estimate with bimanual exam and passage of largest dilator immediately prior to procedure
Total Procedure Time | Measured at clinic visit and on OR day, over 2 day period
  All time required by patient (time in clinic for cervical preparation procedures)
Difficulty of Procedure, as reported by clinician | Measured within 5 minutes after procedure
  Using Visual Analogue Scale (VAS)
Complications/Adverse Events | Intraoperatively
  Estimated blood loss, uterine injury, infection, retained products of conception
Pain Perceived by Patient | Intraoperatively "Measured during dilator placement"
  Using Visual Analogue Scale (VAS)
Overall Patient Experience | Measured post-operatively (30 minutes prior to discharge)
  Using Visual Analogue Scale (VAS)

CONTACTS AND LOCATIONS:
Overall Officials: Principal Investigator, Principal Investigator — Stanford University
Locations (1):
- Planned Parenthood Mar Monte, San Jose, California, United States